CLINICAL TRIAL: NCT07335822
Title: The Effectiveness of Low-Level Laser Therapy in the Treatment of Meralgia Paresthetica
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Merve Sade Dağdeviren, Medical Doctor, Istanbul Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21/02/2025;2011-KAEK-50;37
Record Dates: First submitted 2025-11-28; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-11

CONDITIONS: Meralgia Paresthetica; Lateral Femoral Cutaneous Nerve Entrapment
Keywords: Meralgia Paresthetica; Lateral Femoral Cutaneous Nerve; Entrapment neuropathy; Low-Level Laser Therapy; thigh pain
MeSH Terms: conditions — Femoral Neuropathy; Charcot-Marie-Tooth Disease | interventions — Transcutaneous Electric Nerve Stimulation; Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided into two groups; the first group will receive low-level laser therapy and TENS, while the second group will receive sham laser and TENS therapy.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients in the first group will receive low-level laser therapy, while patients in the second group will receive sham low-level laser therapy. Participants will not be informed about which group they are in. In addition, the outcome assessors will also conduct their assessments blinded to the groups to which the patients belong.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: LOW LEVER LASER THERAPY AND TENS (Active Comparator): Low-level laser therapy will be applied perpendicularly at four different points, delivering a total of 4 J of energy over 12 minutes. TENS electrodes will be placed on the painful anterolateral thigh region
  Interventions: Other: Transcutaneous Electrical Nerve Stimulation (TENS); Other: Low-Level Laser Therapy
- Group 2: SHAM LASER AND TENS THERAPY (Sham Comparator): Sham laser will be applied using the same device and in the same manner; however, no laser beam will be emitted to the designated areas. TENS electrodes will be placed on the painful anterolateral thigh region
  Interventions: Other: Transcutaneous Electrical Nerve Stimulation (TENS)

INTERVENTIONS:
Other: Transcutaneous Electrical Nerve Stimulation (TENS) — TENS electrodes will be placed on the painful anterolateral thigh region in both groups. The stimulation pulse frequency will be set to 100 Hz, and the pulse width will be set to 100 ms.
Other: Low-Level Laser Therapy — Low-level laser therapy will be applied perpendicularly, consistent with the lateral femoral cutaneous nerve projection, delivering a total of 4 J of energy over 12 minutes.
  Arms: Group 1: LOW LEVER LASER THERAPY AND TENS

SUMMARY:
Patients diagnosed with meralgia paresthetica via electromyography (EMG), who present with neuropathic complaints on the lateral thigh to the Physical Medicine and Rehabilitation outpatient clinics of our hospital, will be included in the study after reviewing exclusion criteria. Patients will be randomized into two equal groups using a sealed-envelope system. The treatment group will receive low-level laser therapy (LLLT) combined with simultaneous transcutaneous electrical nerve stimulation (TENS), while the control group will receive placebo laser therapy combined with simultaneous TENS.

An LED gallium-aluminum-arsenide (Ga-Al-As) diode laser device with a power of 1.6 W and a wavelength of 808 nm will be used in the study. The treatment will consist of 10 sessions, applied over two weeks, five days per week.

Demographic data (age, gender, body mass index, and occupation) of all patients included in the study will be recorded. Pain and functional impairment will be evaluated using the VAS, SF-36, PSQI, and S-LANSS scales for all patients. VAS, SF-36, PSQI, and S-LANSS scores will be assessed at the end of the treatment and on the 30th day after treatment completion (6th-week after baseline). The effectiveness of low-level laser therapy will be investigated using statistical data analysis methods.

Low-level laser therapy will be applied perpendicularly, consistent with the lateral femoral cutaneous nerve projection, delivering a total of 4 J of energy over 12 minutes. TENS electrodes will be placed on the painful anterolateral thigh region in both groups. The stimulation pulse frequency will be set to 100 Hz, and the pulse width will be set to 100 ms. In the control group, sham laser will be applied using the same device and in the same manner; however, no laser beam will be emitted to the designated areas.

ELIGIBILITY:
Inclusion Criteria: Patients aged 18 to 70 with neuropathic complaints in the anterolateral thigh, whose diagnosis has been confirmed by sensory conduction studies of the lateral femoral cutaneous nerve.

Exclusion Criteria: - Patients with diabetes mellitus

* Patients with polyneuropathy
* Patients with radicular pain
* Patients receiving treatment for neuropathic pain
* Patients who have received an injection to the lateral femoral cutaneous nerve within the last three months
* Patients who have undergone physical therapy modalities for a diagnosis of meralgia paresthetica within the last three months
* Patients with a history of pelvic surgery
* Patients diagnosed with rheumatologic diseases
* Pregnant women
* Patients with active skin infections
* Malignancy
* Fibromyalgia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Pain will be assessed with Visual Analog Scale. | It will be evaluated at the baseline, at the end of treatment, and at the sixth-week follow-up.
  Visual Analog Scale (VAS) score ranges from 0 to 10. High scores describe more pain, and low scores describe less pain.

SECONDARY OUTCOMES:
Neuropathic pain will be assessed using the S-LANSS scale. | It will be evaluated at the baseline, two weeks after the treatment started, and in the sixth week after the start of the treatment.
  In the S-LANSS pain score, the patient evaluates the worst pain they experienced during the past week. The questions are answered with either 'yes' or 'no.' The total score ranges from 0 to 24. If the total score is twelve or higher, the pain is considered primarily neuropathic in nature.
General health status will be assessed with Short Form 36. | It will be evaluated at the baseline, two weeks after the treatment started, and in the sixth week after the start of the treatment.
  Short Form 36 (SF-36) is a 36-item patient-reported questionnaire that covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). | It will be evaluated at the baseline, two weeks after the treatment started, and in the sixth week after the start of the treatment.
  Consisting of 19 items, the PSQI measures several different aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction.
  Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Fatih, Turkey (Türkiye)